CLINICAL TRIAL: NCT07316257
Title: Value of Adding T2mapping Sequence to Routine MRI Protocol in Assessment of Knee Articular Cartilage in Early Osteoarthritis
Brief Title: Value of Adding T2 Mapping Routine MRI in Assessment of Knee Articular Cartilage Early Osteoarthritis
Acronym: T2 mapping OS
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shrouk Mohamed Gad, DR, Assiut University
Other Study IDs: T2 mapping in osteoarthritis
Record Dates: First submitted 2025-12-16; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Osteearthritis; OA; OA Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MRI — Device that use coil to image asses the articular cartilage of the knee

SUMMARY:
This work aims at elucidating the role of MRI complementary T2 mapping in assessment of the articular knee cartilage for improving sensitivity of detection of early stage of osteoarthritis

DETAILED DESCRIPTION:
Osteoarthritis (OA) is one of the most common degenerative joint diseases, affecting more than 500 million people worldwide (1), causing joint pain and stiffness, and negatively affecting quality of life . The knee is the most commonly affected joint, followed by the hand and hip (1).

It is important clinically to diagnose osteoarthritis in its early stages to prevent its inevitable progression (2) Routine MR imaging sequences used in the identification of knee osteoarthritis can assess articular cartilage morphology, but despite its accuracy for identifying deep hyaline cartilage defects which are considered irreversible cartilage degeneration with limited treatment options, it lacks sufficient sensitivity for early cartilage changes and low-grade chondral lesions which are the reversible stages for the potential alteration of the osteoarthritis progression(2).

T2 mapping of hyaline cartilage is an imaging technique for the qualitative and quantitative detection of the cartilage providing convincing color mapping and quantitative detection of the cartilage mainly regarding architecture and changes in water content, proteoglycan, and collagen matrix ultra-structure associated with early cartilage degeneration(3).

T2 mapping is a time constant describing the rate at which energy transfer occurs between water protons in a magnetic field (spin-spin interactions), leading to signal dephasing. In normal healthy articular cartilage, water protons are largely bound in place by a well-organized matrix of collagen fibers, allowing for rapid dephasing, and therefore low T2 values are seen(4). However, in osteoarthritic articular cartilage, the collagen fibers become disorganized, and there are more mobile water protons, resulting in high T2 values. (4).

ELIGIBILITY:
Inclusion Criteria:

* patients with clinical evidence of osteoarthritis

Exclusion Criteria:

* • contraindications for MRI such as claustrophobia, heart pacemaker and ferromagnetic implants

  * patients in which the misaligned images or distortions due to motion artifacts made the interpretation of the MRI unreliable.
  * Patients with previous knee operation

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: any patient with knee pain with no history of previous lustrophobiaoperation and has no metallic element inside his body with no ca
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-12 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
This work aims at elucidating the role of MRI complementary T2 mapping to measure the changes in T2 relaxation time of the articular knee cartilage in healthy group which there number will be 28 and pateints with early osteoarthritis there number 28 | baseline
  to detect the value of adding T2 mapping to routine MRI in assessment of the articular cartilage in knee osteoarthritis

SECONDARY OUTCOMES:
This work aims at quantitive stratification of osteoarthrtic changes and its impact on treatement | baseline
  to detect the value of adding T2 mapping to routine MRI in assessment of knee articular cartilage in knee osteoarthritis

CONTACTS AND LOCATIONS:
Overall Officials: Abeer Houssein Ali, prof.dr, Study Director — Assiut University; Ahmed Moustafa Mohamed, prof, Study Director — Assiut University

REFERENCES:
- [Background] Le J, Peng Q, Sperling K. Biochemical magnetic resonance imaging of knee articular cartilage: T1rho and T2 mapping as cartilage degeneration biomarkers. Ann N Y Acad Sci. 2016 Nov;1383(1):34-42. doi: 10.1111/nyas.13189. Epub 2016 Jul 29. PMID 27472534
- [Background] Gao S, Peng C, Wang G, Deng C, Zhang Z, Liu X. Cartilage T2 mapping-based radiomics in knee osteoarthritis research: Status, progress and future outlook. Eur J Radiol. 2024 Dec;181:111826. doi: 10.1016/j.ejrad.2024.111826. Epub 2024 Nov 8. PMID 39522425